CLINICAL TRIAL: NCT04222348
Title: Efficacy of Metformin Treatment in Not Controlled With Diet Gestational Diabetes Versus Use of Insulin Therapy
Brief Title: MeDiGes Study: Metformine Use in Gestational Diabetes
Acronym: FIMMET201501
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIM-MET-2015-01
Record Dates: First submitted 2019-12-03; First posted 2020-01-10 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2019-12

CONDITIONS: Diabetes, Gestational; Perinatal Disorder; Puerperal Disorder
MeSH Terms: conditions — Diabetes, Gestational; Puerperal Disorders | interventions — Metformin; Insulin Detemir

STUDY DESIGN:
Intervention Model Description: Inferiority, randomized, open, parallel arms, multicenter clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): 850-2550 mg every 24h.
  Interventions: Drug: Metformin; Drug: Insulin Detemir
- Insulin Detemir (Active Comparator): Individual doses according to glycemic controls.
  Interventions: Drug: Metformin; Drug: Insulin Detemir

INTERVENTIONS:
Drug: Metformin — 850-2550 mg every 24h.
Drug: Insulin Detemir — Insulin detemir associated or not with rapid insulin analogue (aspart) according to individual glycemic controls.

SUMMARY:
Women with gestational diabete (GD) who do not meet glycemic control objectives with diet will be assigned to two treatment groups randomly. One: metformin at a dose of 850-2550mg every 24h; two: insulin detemir associated or not with rapid insulin analogue (aspart) according to your glycemic controls. The Metformin group may additionally receive insulin in a second time in case the glycemic control is not appropriate with monotherapy.

DETAILED DESCRIPTION:
Women with gestational diabete (GD) who do not meet glycemic control objectives with diet will be assigned to two treatment groups randomly. One: metformin at a dose of 850-2550mg every 24h; two: insulin detemir associated or not with rapid insulin analogue (aspart) according to your glycemic controls. The Metformin group may additionally receive insulin in a second time in case the glycemic control is not appropriate with monotherapy.

The objectives are: Demonstrate that treatment with metformin in women with GD (not controlled with diet) can get no lower obstetric and perinatal outcomes than those with standard treatment with insulin.

Demonstrate that glycemic control with metformin in properly selected women, can be equivalent to that obtained with insulin.

ELIGIBILITY:
Inclusion Criteria:

1. 18-45 years old.
2. Diagnosis of GD, with fasting glucose <120 mg / dL.
3. not controlled by diet: fasting capillary blood glucose> 95 mg / dl in at least 2-3 times or 1 hour postprandial >140 mg / dl on, at least 2-3 times a week.
4. 2nd or 3rd trimesters of pregnancy.
5. Able to give informed consent.

Exclusion Criteria:

1. Psychopathological situations that do not guarantee proper adhesion to follow up
2. 1st trimester of pregnancy
3. gastrointestinal diseases that may cause poorer tolerance or increased symptoms with metformin.
4. Patients who can not attend the scheduled consultation.
5. Language barrier limiting for understanding treatment settings
6. Twin pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2020-05-28 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Metformin benefits | 50 weeks
  Change of Weigth
Good glycemic control | 50 weeks
  Change of glycemic levels
Baby wellness | Delivery
  Weight

SECONDARY OUTCOMES:
Adverse event profile | 50 weeks
  Number of adverse events
Fructosamine as a marker of insulinization | 50 weeks
  Concentration of fructosamine
Satisfaction with the treatment | 50 weeks
  Questionnaire of satisfaction with the treatment. Range: 5 (worst)-16 (best)
IL-6 profile | 50 weeks
  IL-6 levels
IL-10 profile and oxidativge stress as well as in lipid profile | 50 weeks
  IL-10 (ultrasensitive PCR) levels
Leptin profile | 50 weeks
  Leptin levels
Ladiponectin and oxidativge stress as well as in lipid profile | 50 weeks
  Ladiponectin levels
LPS profile | 50 weeks
  LPS levels
LBP profile and oxidativge stress as well as in lipid profile | 50 weeks
  LBP levels

IPD SHARING:
Plan to Share IPD: No